CLINICAL TRIAL: NCT07217470
Title: A Pilot Clinical Study to Assess the Correlation Between Fluid Removal During Dialysis and HemoCept Device Data
Brief Title: Fluid Status of ESRD Patients Undergoing Dialysis
Status: Completed | Type: Observational
Sponsor: HemoCept Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRT-017
Record Dates: First submitted 2025-09-16; First posted 2025-10-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: ESRD (End Stage Renal Disease)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The pilot clinical study will assess the correlation between fluid removal during dialysis and HemoCept device data.

ELIGIBILITY:
Inclusion Criteria:

* Subject or representatives must have voluntarily signed the informed consent form before any study related procedures
* Subjects can be any gender, but must be between (and including) 18 and 75 years of age
* Subject has been on dialysis for more than 90 days and has been diagnosed with end stage kidney disease
* Subject is able and willing to provide informed consent and HIPAA authorization.
* Subject is able and willing to meet all study requirements
* Subject is able to place electrodes on bilateral deltoids and above the pant line on the waist.

Exclusion Criteria:

* Subject is pregnant, breast-feeding, or intends to become pregnant during the course of the study.
* Subject has a personal medical history that includes: Long Q-T syndrome, Cardiac channelopathies, genetic heart defects, Seizures, Acute untreated blood clotting disorders or acute untreated bleeding disorders
* Subject has had a heart transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects between (and including) the ages of 18 and 75 and who meet all the Inclusion/Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Correlation between dry weight changes and HemoCept device measurements. | Before and after one dialysis session, over the course of 1 day
  The primary analysis will be conducted using HemoCept device readings taken before dialysis and at the end of dialysis, just prior to return of blood and fluid from the machine. The device data will then be assessed for its comparison to dry weight changes.

SECONDARY OUTCOMES:
Device related adverse events, and the possible correlation of skin tone to device results. | Before and after 1 dialysis session, over the course of 1 day.
  -Device-related adverse events: device-related adverse events included all adverse eventsclassified as definitely, probably, possibly, or undetermined relation to the device or procedure
  --Exploratory correlation of skin tone and device performance: Monk Skin Tone data will be collected to explore potential correlation between subject skin tone and HemoCept device readings.

CONTACTS AND LOCATIONS:
Overall Officials: Jusmin Patel, MD, Principal Investigator — Sierra Nevada Specialty Care
Locations (1):
- Sierra Nevad Specialty Care, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available